CLINICAL TRIAL: NCT06027541
Title: Prospective Research of Young Patients With Early Breast Cancer
Brief Title: Young Patients With Early Breast Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: YEBC
Record Dates: First submitted 2023-01-11; First posted 2023-09-07 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer Female
Keywords: young patients
MeSH Terms: interventions — Surgical Procedures, Operative; Drug Therapy; Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — breast cancer tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: operation — operation methods: breast-conserving surgery, mastectomy, axillary lymph node dissection, sentinal lymphnodes biopsy; chemotherapy regimens: AC, TC, AC-T/P, TCrb, TAC, capecitabine; ovarian protection:GnRHa; endocrine therapy: Aromatase inhibitor, GnRHa, TAM, Fulvestrant, CDK4/6 inhibitors; target therapy: trastuzumab，patuzumab, Pyrotinib.
  Other Names: chemotherapy; radiotherapy; endocrine therapy; targeted therapy; ovarian protection

SUMMARY:
The prognosis of young patients with breast cancer is relatively poor. Chemotherapy damages ovarian function. Endocrine treatment for up to 10 years delays the childbearing time of patients. Treatment regimens in young breast cancer patients are still controversial in the following: 1. Exemption from chemotherapy based on gene prediction results; 2. Removing drugs that damage ovarian function from chemotherapy regimens; 3. Giving ovarian protection drugs during chemotherapy for patients with hormone receptor (HR)+; 4. The right time to get pregnant. In view of the above problems, the treatment scheme recommended in the guidelines cannot meet the personalized needs of young breast cancer patients. The project plans to establish a prognosis model for young patients with breast cancer, and provide the patients hierarchical and refined management, which is significant for prolonging survival time, improving quality of life, and protecting fertility. This project plans to observe the relationship between the characteristics of immune genes, pathological staging, molecular typing, treatment plans and prognosis in the cohort of young breast cancer patients, and establish a young breast cancer prognosis model and verify it. The project is expected to establish a prognosis model and provide a hierarchical and personalized precision treatment plan for young breast cancer patients, so as to prolong the survival time, improve the fertility rate, and improve the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* patients with breast cancer received operation in Peking Union Medical College Hospital
* age ≤40 year old and ≥20 years old
* treatment regimen was made in Peking Union Medical College Hospital

Exclusion Criteria:

* patients without pathological information
* patients with metastasis
* patients with history of other malignant tumor (except for completely cured cervical carcinoma in situ or basal cell carcinoma or squamous cell skin carcinoma)
* patients with palliative resection of breast

Max Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients with breast cancer receiving operation in Peking Union Medical College Hospital
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
5-year disease free survival (DFS) | 5 year
  DFS: From the time of surgery to the time of recurrence or metastasis, calculated on a monthly basis, until the most recent discovery of recurrence or metastasis.

SECONDARY OUTCOMES:
5-year overall survival (OS) | 5-year
  OS: From the time of surgery to death from any cause, calculated on a monthly basis.
5-year recurrence | 5-year
  Recurrence: Recurrence in the ipsilateral breast, axillary, or supraclavicular lymph nodes comfired by pathological biopsy confirmation.
5-year metastasis | 5-year
  Metastasis: metastasis was detected by CT, MRI, nuclide scanning or ultrasound in liver, lung, bone, brain, and other areas, without being confirmed by pathology.
the correlation between poor characteristics and survival | 5-year
  clinical characteristics': T stage, N stage, tumor grade, age group, with or without ovaian protection, with or without chemotherapy/radiotherapy, operation method.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China